CLINICAL TRIAL: NCT00914641
Title: A Randomized, Open-Label, Single Dose, Four Way Cross-Over Bioavailability Study Comparing Three Modified Release Formulations Of Apixaban Tablets To Apixaban Immediate Release Tablets In Healthy Volunteers
Brief Title: Bioavailability Study Comparing Modified Release To Immediate Release Apixaban Tablets In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B0661007; CV185071
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Thrombosis
Keywords: formulation; sustained release; modified release; extended release
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apixaban Cross-over (Other)
  Interventions: Drug: Apixaban IR; Drug: Apixaban MR1; Drug: Apixaban MR2; Drug: Apixaban MR3

INTERVENTIONS:
Drug: Apixaban IR — immediate release tablet, 10 mg, single dose
Drug: Apixaban MR1 — modified release tablet 1, 10 mg, single dose
Drug: Apixaban MR2 — modified release tablet 2, 10 mg, single dose
Drug: Apixaban MR3 — modified release tablet 3, 10 mg, single dose

SUMMARY:
To estimate the pharmacokinetics of apixaban when administered as three different modified release formulation tablets relative to that when apixaban is administered as an immediate release tablet

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female patients
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* History or evidence of abnormal bleeding or clotting disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Apixaban PK: Cmax, C24, AUClast, AUCinf, Tmax, and half-life (t½) | 96 hours
Safety and tolerability as determined by adverse event reporting, clinical laboratory results, vital signs, physical examinations, and ECGs. | per treatment period of 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0661007&StudyName=Bioavailability%20Study%20Comparing%20Modified%20Release%20To%20Immediate%20Release%20Apixaban%20Tablets%20In%20Healthy%20Volunteers